CLINICAL TRIAL: NCT07005583
Title: Clinical Study of QL1706 in Combination With Olaparib for the Treatment of Patients With Previously Treated Homologous Recombination Repair-Deficient Recurrent or Metastatic Triple-Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20250403
Record Dates: First submitted 2025-05-12; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Triple-Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 + Olaparib (Experimental)
  Interventions: Drug: QL1706 Plus Olaparib

INTERVENTIONS:
Drug: QL1706 Plus Olaparib — QL1706: 5 mg/kg administered via intravenous (IV) infusion every 3 weeks (Q3W). Olaparib: 300 mg (two 150 mg tablets) taken orally twice daily (BID). Treatment will continue until protocol-defined discontinuation criteria are met, including disease progression, unacceptable toxicity, withdrawal of consent, or death.

SUMMARY:
This is a single-arm, prospective, Phase II clinical trial designed to assess the efficacy and safety of QL1706 in combination with olaparib in patients with recurrent or metastatic triple-negative breast cancer (TNBC) harboring homologous recombination repair deficiency (HRD) who have received prior therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and comply with the requirements of this study, and voluntarily sign the informed consent form.
2. Female breast cancer patients aged ≥18 and ≤75 years, with histologically or cytologically confirmed recurrent or metastatic triple-negative breast cancer (TNBC) as defined by the latest ASCO/CAP guidelines (based on the most recent biopsy or other pathological specimens).
3. Have received at least 1 but no more than 2 prior lines of anti-tumor therapy （ Disease progression during or within 12 months after completing neoadjuvant/adjuvant therapy counts as one line of therapy；Must have received taxane-based therapy at any stage；A maximum of 1 prior antibody-drug conjugate (ADC) therapy is allowed.）
4. Documented homologous recombination repair deficiency (HRD) (BRCA1/2 mutation and/or HRD-positive status.
5. Any PD-L1 expression status (no restriction).
6. Have at least one measurable lesion according to RECIST 1.1 criteria (assessed by CT or MRI). Bone-only lesions are considered non-measurable and do not qualify for enrollment.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
8. Availability of tumor tissue samples for biomarker testing.
9. Ability to swallow tablets normally.
10. Expected survival ≥3 months.
11. Presence of adequate bone marrow and organ function.

Exclusion Criteria:

1. Prior treatment with immune checkpoint inhibitors (e.g., anti-PD-1/PD-L1, anti-CTLA-4) or PARP inhibitors (e.g., olaparib, niraparib).
2. Current use of immunosuppressive agents or systemic corticosteroids for immunosuppressive purposes (>10 mg/day prednisone or equivalent) within 2 weeks prior to enrollment.
3. History of severe allergic reactions to monoclonal antibodies.
4. Discontinuation of prior anti-PD-1/PD-L1/CTLA-4 therapy due to immune-related toxicity.
5. Known history or evidence of interstitial lung disease or active non-infectious pneumonitis.
6. History of CNS metastases or current CNS metastases. Baseline imaging to confirm absence of brain metastases is not mandatory. Patients with unknown CNS status but clinical signs suggestive of CNS involvement are eligible if CNS metastases are ruled out by CT/MRI.
7. History of other malignancies (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless disease-free for ≥3 years.
8. Uncontrolled hypertension (SBP ≥140 mmHg or DBP ≥90 mmHg) despite antihypertensive therapy. History of hypertensive crisis or hypertensive encephalopathy.
9. History of unstable angina, myocardial infarction, chronic heart failure (LVEF <50%), or clinically significant arrhythmias requiring treatment (except stable atrial fibrillation) within 6 months prior to treatment.
10. Current therapeutic anticoagulation or thrombolysis (prophylactic low-dose aspirin/LMWH permitted).
11. Clinically significant effusions (pleural, peritoneal, or pericardial) requiring drainage, unless stabilized post-drainage per investigator assessment.
12. Arterial/venous thromboembolic events (e.g., CVA, TIA, DVT, PE) within 6 months prior to enrollment.
13. Major vascular disease (e.g., aortic aneurysm requiring repair or recent peripheral arterial thrombosis) within 6 months.
14. Major surgery within 4 weeks prior to treatment or anticipated during the study (excluding diagnostic procedures).
15. Urine protein ≥++ on dipstick with confirmed 24-hour urine protein >1.0 g.
16. Prior radiotherapy (except palliative bone radiation), chemotherapy, or surgery (excluding biopsy) within 4 weeks before treatment initiation; <4 weeks since last antibody therapy; <5 half-lives since last targeted therapy (including investigational agents); or unresolved toxicities (>CTCAE grade 1, except alopecia).
17. Active infection, unexplained fever ≥38.5°C within 7 days, or baseline WBC >15×10⁹/L.
18. Immunodeficiency (e.g., HIV); HBsAg-positive with HBV DNA ≥2000 IU/mL; or HCV antibody-positive.
19. Active or history of autoimmune diseases (e.g., autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism). Exceptions: vitiligo, childhood asthma resolved without intervention, or stable hypothyroidism on hormone replacement.
20. Live vaccination within 4 weeks prior to treatment or planned during the study.
21. Planning pregnancy, pregnancy, or suckling period;
22. The investigator judged that the patients are not suitable for participating in this trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2030-05-20 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) - investigator assessment | Up to 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) - Investigator assessment | Up to 2 years
Duration of response (DOR) - Investigator assessment | Up to 2 years
Overall survival (OS) | Up to 5 years
Number of participants with adverse events (AEs), Serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs) | Up to 5 years

OTHER OUTCOMES:
Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1% | Up to 2 years
  PFS was determined in participants who had a PD-L1 CPS of ≥1% as measured by immunohistochemistry assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No